CLINICAL TRIAL: NCT05547880
Title: CNS Correlates of Extended Sleep Restriction
Status: Completed | Type: Observational
Sponsor: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Intrepid Center of Excellence (U.S. Federal Agency)
Responsible Party: Principal Investigator, Samantha Riedy, Principal Investigator, Walter Reed Army Institute of Research (WRAIR)
Other Study IDs: 2804; MO220146 (Other Grant/Funding Number: Military Operational Medicine Research Program)
Record Dates: First submitted 2022-07-26; First posted 2022-09-21 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Sleep Restriction
Keywords: Sleep Restriction; Alertness; Performance; Neuroinflammation; Biomarker
MeSH Terms: conditions — Neuroinflammatory Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: [11C]ER176 — Brain PET with [11C]ER176. [11C]ER176 is a PET ligand that images TSPO.

SUMMARY:
Chronic sleep restriction is ubiquitous in both the general population and the military. The deleterious effects of sleep loss on human alertness and cognitive performance have been documented in numerous studies dating back to the nineteenth century. Over the past decade, evidence has emerged indicating that chronic sleep restriction may also precipitate deleterious, long lasting neuropathological changes in the brain. The purpose of this study is to determine neuropathological effects of sleep restriction and identify physiological mechanisms that correlate with sleep loss-induced performance impairment.

ELIGIBILITY:
* Ages 18 to 39 (inclusive)
* A body mass index (BMI) below 30.
* Weigh at least 140 lbs
* Females must not be pregnant or nursing, and must be on some form of birth control, if sexually active (e.g., oral contraceptive, condom, intrauterine device, etc.)
* No history of sleeping problems such as insomnia or sleep apnea.
* Test negative for alcohol, nicotine, illegal drugs, and not take certain medications.
* Must not excessively consume alcohol or caffeine.
* Active duty and Federal employees must be on leave during participation.
* No history of heart disease (high blood pressure), neurologic disorder (such as seizures of epilepsy), liver disease, kidney disease, or metabolic disorder or diabetes.
* No history of underlying acute or chronic pulmonary disease requiring daily inhaler use.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Positron Emission Tomography (PET) based measurement of neuroinflammation | 3 Days
  Positron Emission Tomography (PET) is the brain imaging method and [11C]ER176 is the PET radioligand providing an index of neuroinflammation

SECONDARY OUTCOMES:
Psychomotor Vigilance Task (PVT) | 55 Days
  Measure of cognitive performance
Actigraphy | 55 Days
  Activity monitoring used to infer sleep-wake patterns
Polysomnographic measurements of sleep and wakefulness | 19 Days
  Measure of various aspects of sleep and wakefulness

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed Army Institute of Research, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belenky G, Wesensten NJ, Thorne DR, Thomas ML, Sing HC, Redmond DP, Russo MB, Balkin TJ. Patterns of performance degradation and restoration during sleep restriction and subsequent recovery: a sleep dose-response study. J Sleep Res. 2003 Mar;12(1):1-12. doi: 10.1046/j.1365-2869.2003.00337.x. PMID 12603781

DOCUMENTS (1):
  • Informed Consent Form (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT05547880/ICF_000.pdf